CLINICAL TRIAL: NCT01466101
Title: Analgesic Effect of Pregabalin in Patients Undergoing Total Abdominal Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution. No subjects screened or enrolled.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christian Altman, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00025229
Record Dates: First submitted 2010-04-20; First posted 2011-11-07 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Pain
Keywords: Hysterectomy; Pain; Pregabalin
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin administration (Active Comparator): Administration of pregabalin
  Interventions: Drug: Pregabalin administration
- Placebo (Placebo Comparator): Administration of placebo
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Placebo administration — Administration of placebo
  Arms: Placebo
Drug: Pregabalin administration — Administration of pregabalin
  Arms: Pregabalin administration

SUMMARY:
Pregabalin will decrease the total amount of opioid required in patients undergoing total abdominal hysterectomy. In addition, pregabalin will decrease the incidence of opioid-related side effects in patients undergoing total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1-2
* Age 18-64
* BMI 18-35
* Scheduled for elective total abdominal hysterectomy (with or without bilateral salpingo-oophorectomy)
* Gender: Female
* Consent: Obtained

Exclusion Criteria:

* Patient refusal
* Allergy to study medication(s)
* Preoperative use of gabapentinoids
* Preoperative use of anticonvulsants
* Daily use of analgesics
* Hepatic disease
* Renal insufficiency (Cr >2.0)
* Alcohol or drug abuse
* Pregnancy
* Language: Non-English speaking
* Patient expected to remain intubated after procedure

Dropout:

* Patient request
* Surgeon request
* Allergic reaction to pregabalin
* Surgical procedure significantly altered from scheduled procedure

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01

PRIMARY OUTCOMES:
total hydromorphone consumption | 24 hours
  total hydromorphone consumption 24 hours post operatively

SECONDARY OUTCOMES:
Pain Scores postoperative | Post operative period
  Post operative pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Christian Altman, MD, Principal Investigator — Northwestern University

REFERENCES:
- [Background] Joshi GP. Multimodal analgesia techniques and postoperative rehabilitation. Anesthesiol Clin North Am. 2005 Mar;23(1):185-202. doi: 10.1016/j.atc.2004.11.010. PMID 15763418
- [Background] Tang R, Evans H, Chaput A, Kim C. Multimodal analgesia for hip arthroplasty. Orthop Clin North Am. 2009 Jul;40(3):377-87. doi: 10.1016/j.ocl.2009.04.001. PMID 19576406
- [Background] Gilron I. Gabapentin and pregabalin for chronic neuropathic and early postsurgical pain: current evidence and future directions. Curr Opin Anaesthesiol. 2007 Oct;20(5):456-72. doi: 10.1097/ACO.0b013e3282effaa7. PMID 17873599
- [Background] Turan A, Karamanlioglu B, Memis D, Usar P, Pamukcu Z, Ture M. The analgesic effects of gabapentin after total abdominal hysterectomy. Anesth Analg. 2004 May;98(5):1370-3, table of contents. doi: 10.1213/01.ane.0000108964.70485.b2. PMID 15105217
- [Background] Gilron I, Orr E, Tu D, O'Neill JP, Zamora JE, Bell AC. A placebo-controlled randomized clinical trial of perioperative administration of gabapentin, rofecoxib and their combination for spontaneous and movement-evoked pain after abdominal hysterectomy. Pain. 2005 Jan;113(1-2):191-200. doi: 10.1016/j.pain.2004.10.008. PMID 15621380
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. Premedication with pregabalin 75 or 150 mg with ibuprofen to control pain after day-case gynaecological laparoscopic surgery. Br J Anaesth. 2008 Jun;100(6):834-40. doi: 10.1093/bja/aen098. Epub 2008 Apr 29. PMID 18448418
- [Background] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Background] Cabrera Schulmeyer MC, de la Maza J, Ovalle C, Farias C, Vives I. Analgesic effects of a single preoperative dose of pregabalin after laparoscopic sleeve gastrectomy. Obes Surg. 2010 Dec;20(12):1678-81. doi: 10.1007/s11695-009-9944-1. Epub 2009 Aug 29. PMID 19727980
- [Background] Brandsborg B, Nikolajsen L, Hansen CT, Kehlet H, Jensen TS. Risk factors for chronic pain after hysterectomy: a nationwide questionnaire and database study. Anesthesiology. 2007 May;106(5):1003-12. doi: 10.1097/01.anes.0000265161.39932.e8. PMID 17457133